CLINICAL TRIAL: NCT05157685
Title: Evaluation of the Efficacy of 3-month Continuous Extended Treatment With Azithromycin in Idiopathic Purulent Oedematous Sinusitis in Adults: a Multicentre Randomised Controlled Trial
Brief Title: Evaluation of the Efficacy of Azithromycin in Idiopathic Purulent Oedematous Sinusitis in Adults
Acronym: SOPAZITHRO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOPAZITHRO; 2020-001227-13 (EudraCT Number)
Record Dates: First submitted 2021-10-28; First posted 2021-12-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Sinusitis, Chronic; Sinus Infection Chronic
MeSH Terms: conditions — Sinusitis; Bronchiolitis Obliterans Syndrome | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin oral tablet (Experimental): Azithromycin 250 mg once daily morning or evening (with or without meals)
  Interventions: Drug: Azithromycin Oral Tablet
- Placebo (Placebo Comparator): Placebo once daily morning or evening (with or without meals)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin Oral Tablet — Treatment assigned by randomization will be prescribed immediately. The active or placebo will be dispensed by the centre's pharmacy. Treatment will be taken in the morning or evening for 3 months.
  Other Names: active arm
  Arms: Azithromycin oral tablet
Drug: Placebo — Treatment assigned by randomization will be prescribed immediately. The active or placebo will be dispensed by the centre's pharmacy. Treatment will be taken in the morning or evening for 3 months.
  Other Names: comparator arm
  Arms: Placebo

SUMMARY:
Purulent Oedematous Sinusitis (POS) is a particular form of chronic rhinosinusitis observed in 2% of the general population. In spite of its heavy impact on the quality of life, There is no established recommendation for the treatment of primary POS. Long-term low-dose macrolides are currently proposed for these forms of chronic rhinosinusitis when conventional treatments (local corticosteroids, saline rinsing, iterative short courses of antibiotics targeted on pathogens, and surgical opening and drainage) have failed. This treatment with macrolides is currently applied off-label.

This study aims to assess the efficacy of macrolides in POS. An extensive workup is fulfilled to exclude other forms of chronic rhinosinusitis (Th2 biased inflammatory diseases, allergic diseases) (allergy, nasosinusal polyposis) or those due to cystic fibrosis or immune deficiency.

DETAILED DESCRIPTION:
POS is a particular form of chronic rhinosinusitis described in 2% of the general population. They lead to an alteration in the quality of daily life with a significant impact on the professional life of 70% of patients. They can be of idiopathic or of secondary origin. The most frequent secondary forms are those observed in cystic fibrosis and immune deficiencies. The pathophysiology of primary POS remains poorly understood, involving Th1-type inflammation and various bacteria (with Staphylococcus Aureus in the forefront). Bacteria could impair the ciliary beat, perpetuating infection and mucosal inflammation. There is no established recommendation for the treatment of primary POS Long-term low-dose macrolides are currently proposed for these forms of chronic rhinosinusitis when conventional treatments (local corticosteroids, saline rinsing, iterative short courses of antibiotics adapted to the germs found, and surgical drainage) have failed. This treatment with macrolides is currently used off label.

Macrolides are effective on most gram-positive and gram-positive bacteria. Macrolides also have immunomodulatory properties on the Th1 immune response. This effect is maintained even in the presence of macrolide-resistant bacteria. In chronic obstructive pulmonary disease, daily administration of half-dose macrolides over the long term (HDLT) has been shown to be effective in reducing the frequency of infectious exacerbations. Uncontrolled trials have described an improvement in symptom scores in chronic rhinosinusitis with or without polyps. The results observed in randomized trials versus placebo are contradictory. A meta-analysis published in 2013 based on these 2 randomized studies was inconclusive regarding the efficacy of HDLT macrolides. The heterogeneity of the inclusion criteria with rhinosinusitis of a different proTh-2 inflammatory profile corresponding to that usually observed in nasal polyposis could explain this lack of result. A review of the literature published in 2017 on HDLT macrolides based on 52 publications observed a very wide diversity of antibiotic protocols in terms of the molecule chosen, the administration scheme and the duration of treatment (8 to 24 weeks). The number of patients studied was often small, which affected the statistical power of the results obtained. The authors of this review conclude by stressing the need to conduct placebo-controlled studies on large populations of patients selected on the phenotypic level.

This study propose to evaluate the value of HDLT macrolides in this specific etiological setting. This project plans to exclude all chronic rhinosinusitis of Th2 inflammatory origin (allergy, nasosinusal polyposis) or those due to cystic fibrosis or immune deficiency. In addition, the inclusion centers selected in Ile de France have the necessary expertise to evaluate the impact of azithromycin on mucociliary clearance, notably with the development of innovative tools to measure the efficiency of the ciliary beat (high-speed video microscopy and particle tracking).At the same time, the tolerance of HDLT macrolides measured in patients with cystic fibrosis or chronic obstructive pulmonary disease (COPD) is excellent, provided that the well-documented contraindications are respected. No serious adverse effects have been reported, apart from cases of transient or permanent moderate hearing loss requiring audiometric monitoring.

No specific study regarding the treatment of primary POS is available to date, even tough POS is very prevalent and its management is still associated with poor patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years and less than 70 years of age
* Chronic rhinosinusitis (> 12 weeks of evolution) meeting the definition published in the European Paper Position2012 (1) and corresponding exclusively to the following endoscopic and CT criteria:

  * Nasal endoscopy showing bilateral and diffuse involvement associating edema of the mucosa of the nasal cavities and meatus with the presence of mucopurulent secretions in these areas
  * Nasosinus CT scan showing diffuse and bilateral pansinus opacities involving at least the maxillary sinuses and the anterior and posterior ethmoids
* Persistent intractable purulent rhinosinusitis despite at least 2 antibiotic therapies
* Signed informed consent of the patient
* Membership in a health insurance plan or beneficiary

Exclusion Criteria:

* Pregnancy or breastfeeding
* PCOS of identified primary cause (identified immune deficiency, cystic fibrosis, HIV)
* Chronic non-purulent rhinosinusitis (nasosinusal polyposis, allergic rhinosinusitis)
* Localized chronic suppurative rhinosinusitis (single sinus, unilateral, frontal or maxillary or sphenoidal)
* Severe hepatic insufficiency (factor V level < 50%)
* Severe renal insufficiency (stage 4 (GFR < 30 ml/min/1.73 m2) and/or creatinine < 40 ml/min)
* Severe heart failure (old age, ischemic heart disease, episode of recurrent cardiac arrest; hypotension, NYHA functional stage III-IV; widened QRS, complex ventricular arrhythmias; hyponatremia (Na <135mmol/l); stage 4 renal failure (GFR < 30 ml/min/1.73 m2); severely depressed LVEF (< 30%)
* Documented moderate pre-existing sensorineural hearing loss with a mean pure tone threshold in the poorer ear in bone conduction >30 dB across all 3 frequencies (500, 1000 and 2000 Hz) or in only one ear (unilateral deafness).
* Major cognitive impairment or lack of French language skills preventing completion of SNOT-22 and SF-36 questionnaires
* Patient with galactose intolerance, total lactase deficiency or glucose-galactose malabsorption syndrome (rare hereditary diseases)
* Patient with peanut or soy allergy
* Patient allergic to macrolides
* Patients who are intolerant or allergic to any of the excipients of azithromycin or placebo
* Treatment with azithromycin in the previous 3 months
* Long QT on ECG ((>440ms for male and >450ms for female) or cardiac arrhythmia or bradycardia (<60btm).The calculation of the corrected QT should be carried out using the Bazett formula.
* Hypokalemia or hypomagnesemia on blood ionogram
* Confirmed or suspected atypical mycobacteriosis
* Contraindicated drug combinations with macrolides (K-vitamins or drugs containing cisapride, colchicine, ergotamine or dihydroergotamine)
* Cautionary drug combinations (non-inclusion criteria)

  * Atorvastatin (Increased risk of concentration-dependent rhabdomyolysis-type adverse events due to decreased hepatic metabolism of the cholesterol-lowering drug.
  * Ciclosporin (risk of increased ciclosporin blood levels and creatinine levels)
  * Digoxin (increase in digoxemia due to increased absorption of digoxin), Drugs likely to cause torsades de pointes, in particular class IA (e.g. quinidine) and class III (e.g. amiodarone, sotalol) antiarrhythmics, antipsychotics (e.g. phenothiazines, pimozide), tricyclic antidepressants (e.g. citalopram), certain fluoroquinolones (e.g. moxifloxacin, levofloxacin) (increased risk of ventricular rhythm disturbances)
  * Simvastatin (increased risk of rhabdomyolysis-type adverse effects (concentration-dependent), due to decreased hepatic metabolism of the cholesterol-lowering agent)
  * Ivabradine (increased risk of ventricular rhythm disorders),
  * Hypokalemic drugs
  * Bradycardia drugs
* Patients with severe cholestasis
* Patients under guardianship or curatorship
* Patients with hematologic malignancies who have undergone hematopoietic stem cell transplantation
* History of facial radiotherapy
* History of rhinosinus cancer
* Participation in other category 1 research at the time of inclusion or in the month prior to inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2027-11-21 (Estimated); Study Completion 2027-11-21 (Estimated)

PRIMARY OUTCOMES:
Comparison of sinonasal outcome test (SNOT) 22 | 3 months
  Comparison of the means of the Sinonasal Outcome Test (SNOT 22) specific quality of life scores after 3 months of treatment. (min = 0, max = 110)

SECONDARY OUTCOMES:
Number of infectious rhinosinus exacerbations | 3 months
  The number of infectious rhinosinus exacerbations during the 3-month period,
Number of courses of antibiotics used | 3 months
  Number of courses of antibiotics used during the 3-month period other than azithromycin or placebo
Visual analog scales of symptoms | 6 months
  Visual analog scales (VAS) of symptoms (self-assessment) (nasal obstruction, rhinorrhea, facial pain, smell disorder, nasal hyperactivity, epistaxis). The VAS measures the intensity of pain on a scale from 0 to 10.
Semi-quantitative symptom scale | 6 months
  Semi-quantitative 4-point symptom scale assessed by the practitioner (min = 0, max = 3)
Semi-quantitative nasal endoscopy score | 6 months
  Semi-quantitative nasal endoscopy score (0: absent/1: present) for each of the following items: presence of pus, edema, erythema, crusts, polyps, scored out of 5 per nasal cavity (maximum score of 10) (Lund Kennedy score),
Quantitative Lund MacKay CT score | 6 months
  Quantitative Lund MacKay CT score (0: no sinus opacity, 1: moderate opacity, 2: total opacity) measured on 12 for each side (score of 24 maximum),
Nasal inflammation flow | 6 months
  Nasal inflammation (nasal nitric oxide (NO) flow, neutrophil polynuclear cell (NPC) and lymphocyte infiltrate on nasal cytology and assays of interleukin 6, 8 and elastase produced by NPCs in nasal secretions)
General quality of life | 6 months
  General quality of life Short form 36 (SF-36) (min=1, max=100)
Days off work | 6 months
  Number of days off work in the 3 months prior to treatment and the number of days off work during the 3 months of treatment
Olfactory score | 6 months
  Olfactory score (sniffing's stick test),
Bacteria present on the protected nasal swab | 6 months
  Identification and quantification of bacteria observed on the protected nasal swab (semi-quantitative score
Number of participants with clinical adverse events as assessed by compliance | 3 months
  Clinical tolerance evaluated by the effective intake of tablets
Number of participants with biological adverse events as assessed by compliance | 3 months
  Biological tolerance evaluated by the effective intake of tablets
Residual effect of the treatment using the SNOT 22 quality of life questionnaires | 6 months
  At 6 months (i.e., 3 months after cessation of treatment), the residual effect of treatment will be measured using the SNOT 22 quality of life questionnaires
Residual effect of the treatment using the SF-36 quality of life questionnaires | 6 months
  At 6 months (i.e., 3 months after cessation of treatment), the residual effect of treatment will be measured using the SF-36 quality of life questionnaires
Residual effect of the treatment using the VAS score | 6 months
  At 6 months (i.e., 3 months after cessation of treatment), the residual effect of treatment will be measured using the VAS score. The VAS measures the intensity of pain on a scale from 0 to 10.
Residual effect of the treatment using the semi-quantitative symptom scale | 6 months
  At 6 months (i.e., 3 months after cessation of treatment), the residual effect of treatment will be measured using the semi-quantitative symptom scale
Residual effect of the treatment using the nasal endoscopy | 6 months
  At 6 months (i.e., 3 months after cessation of treatment), the residual effect of treatment will be measured using the nasal endoscopy
Residual effect of the treatment using the bacteriological samples. | 6 months
  At 6 months (i.e., 3 months after cessation of treatment), the residual effect of treatment will be measured using the bacteriological samples.
Quantitative aspect of the ciliary beat | 6 months
  Quantitative aspect of the ciliary beat (frequency of the beat in Hertz) on a small number of centers having the equipment
Qualitative aspect of the ciliary beat | 6 months
  Qualitative aspect of the ciliary beat (coordination (normal or dyskinetic), index of efficiency)) on a small number of centers having the equipment

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Bordeaux, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - CHU Bicêtre, AP-HP, Le Kremlin-Bicêtre
  - CHU Lille, Lille
  - CHU de la Croix Rousse, Lyon
  - Hospices de Lyon, Lyon
  - Hôpitaux Universitaires de Marseille Conception, Marseille
  - CHRU de Nancy, Nancy
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Hôpital Lariboisiere, Paris
  - CHU Cochin, Paris
  - CHU Toulouse, Toulouse
  - Centre Hospitalier Intercommunal, Créteil, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No